CLINICAL TRIAL: NCT00786812
Title: An Open-label, Multicenter Study of Treatment With Nilotinib in Adult Patients With Imatinib - Resistant or - Intolerant Chronic Myeloid Leukemia in Blast Crisis, Accelerated Phase or Chronic Phase
Brief Title: Study of Treatment With Nilotinib in Adult Patients With Imatinib - Resistant or - Intolerant Chronic Myeloid Leukemia in Blast Crisis, Accelerated Phase or Chronic Phase
Acronym: MACS0439
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107ABR03
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Leukemia; adult chronic myeloid leukemia; imatinib; nilotinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia | interventions — nilotinib

ARMS (2):
- CAMN107A2109 Extension Patients (Other)
  Interventions: Drug: Nilotinib
- AMN107 Naive (Other)
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib

SUMMARY:
Maintain and monitor long-term hematological and cytogenetic responses previously obtained by patients participating in the [CAMN107A2109] study

ELIGIBILITY:
Inclusion Criteria:

1. patients currrently participating in Novartis study CAMN107A2109
2. imatinib - resistant or intolerant - Philadelphia chromosome-positive CML in chronic (CML-CP)accelerated phase (CML-AP) or in blast crisis (CML-BC)
3. males or females ≥18 years of age
4. WHO Performance Status of ≤ 2
5. patients must have the following laboratory values: ALT and AST ≤ 2.5 x ULN or ≤ 5.0 x ULN if considered due to tumor

Exclusion Criteria:

1. Impaired cardiac function; use of therapeutic coumarin derivatives
2. patients who have undergone a major surgery and have not recovered from side effects of such therapy within 15 days
3. patients who are pregnant or breast feeding, or adults of reproductive potential not employing an effective method of birth control
4. patients who have received chemotherapy ≤ 1 week or who are within 5 half-lives of their last dose of chemotherapy
5. ,.patients who have received imatinib or dasatinib at least 3 days prior to beginning of study drug or who have not recovered from side effects of such therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2008-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Disease response (complete hematologic response, cytogenetic response) and progression at or until 24 months, depending of the case every 3 months | 3 - 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- Brazil (8):
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Campinas, São Paulo
  - Novartis Investigative Site, Jaú, São Paulo
  - Novartis Investigative Site, Ribeirão Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo